CLINICAL TRIAL: NCT00375375
Title: Effect of Lactulose on Minimal Hepatic Encephalopathy and Health-Related Quality of Life
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minimal hepatic encephalopathy
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2007-03

CONDITIONS: Minimal Hepatic Encephalopathy; Hepatic Encephalopathy
Keywords: Minimal hepatic encephalopathy; Hepatic encephalopathy; Subclinical hepatic encephalopathy; Health related quality of life
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Lactulose

INTERVENTIONS:
Drug: Lactulose

SUMMARY:
Minimal hepatic encephalopathy (MHE) has a negative effect on patients' daily functioning. No study has so far investigated the effect of treatment related improvement in cognitive functions on health related quality-of-life (HRQOL). This study was carried out to determine the influence of treatment on psychomotor performance and on HRQOL in patients with MHE.

The mean number of abnormal NP tests decreased significantly in patients in treated group compared with patients in untreated group MANOVA for time and treatment, P =.001). Mean total SIP score improved among patients in the treated group after 3 months compared with patients in untreated group after 3 months (MANOVA for time and treatment, P=.002). Improvement in HRQOL was related to the improvement in psychometry. In conclusion, treatment with lactulose improves both cognitive functions and HRQOL in cirrhotic patients with MHE.

DETAILED DESCRIPTION:
The study has been published in March 2007 in Hepatology

Lactulose Improves Cognitive Functions and Health-Related Quality of Life in Patients with Cirrhosis WhoHave Minimal Hepatic Encephalopathy.Srinivasa Prasad, Radha K. Dhiman, Ajay Duseja, Yogesh K. Chawla, Arpita Sharma, and Ritesh Agarwal. (HEPATOLOGY 2007;45:549-559.)

ELIGIBILITY:
Inclusion Criteria:

* All the patients diagnosed as having cirrhosis of liver

Exclusion Criteria:

* Overt HE or a history of overt HE;
* History of recent (< 6 weeks) alcohol intake;
* Infection, recent (< 6 weeks) antibiotic use or gastrointestinal bleeding;
* History of recent (< 6 weeks) use of drugs affecting psychometric
* Performances like benzodiazepens, antiepileptics, psychotropic drugs;
* History of shunt surgery or transjugular intrahepatic portosystemic shunt for portal hypertension;
* Electrolyte imbalance;
* Renal impairment;
* Presence of hepatocellular carcinoma;
* Severe medical problems such as congestive heart failure, pulmonary disease, neurological or psychiatric disorder, etc., that could influence quality-of-life measurement;
* Inability to perform NP tests and to complete the SIP questionnaire due to bad vision.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2004-01; Study Completion 2004-12

PRIMARY OUTCOMES:
Improvement in minimal hepatic encephalopathy and health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Radha K Dhiman, MD,DM, FACG, Principal Investigator — Postgraduate Institute of Medical Education and Research, Chandigarh-160012, India
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Uttarakhand, India

REFERENCES:
- [Result] Prasad S, Dhiman RK, Duseja A, Chawla YK, Sharma A, Agarwal R. Lactulose improves cognitive functions and health-related quality of life in patients with cirrhosis who have minimal hepatic encephalopathy. Hepatology. 2007 Mar;45(3):549-59. doi: 10.1002/hep.21533. PMID 17326150